CLINICAL TRIAL: NCT00156910
Title: A Study Using Botulinum Toxin Type A as Headache Prophylaxis for Migraine Patients With Frequent Headaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-079
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-10

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- botulinum toxin Type A (Experimental): Two treatment sessions in the double-blind phase and three treatment sessions in the open-label extension phase. Total minimum dose is 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas with the total maximum dose of 195 U with 39 head/neck injections.
  Interventions: Biological: Botulinum Toxin Type A
- Placebo (saline) (Placebo Comparator): Two treatment sessions in the double-blind phase. Total minimum dose in 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas and the total maximum dose is 195 U with 39 head/neck injections.
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Two treatment sessions in the double-blind phase and three treatment sessions in the open-label extension phase. Total minimum dose is 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas with the total maximum dose of 195 U with 39 head/neck injections.
  Other Names: BOTOX®
  Arms: botulinum toxin Type A
Other: Placebo (saline) — Two treatment sessions in the double-blind phase. Total minimum dose in 155 U with 31 fixed-site, fixed dose injections across seven specific head/neck muscle areas and the total maximum dose is 195 U with 39 head/neck injections.
  Arms: Placebo (saline)

SUMMARY:
This is a 60 week study including a double-blind phase followed by an open-label extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Frequent migraine (>=15 headache days per month)
* >=4 distinct headache episodes lasting >=4 hours
* >=50% of baseline headache days migraine/probable migraine days

Exclusion Criteria:

* Previous use of botulinum toxin of any serotype or immunization to any botulinum toxin serotype
* Any medical condition that puts the patient at increased risk with exposure to BOTOX
* Diagnosis of complicated migraine, chronic tension-type headache, hypnic headache, hemicrania continua, new daily persistent headache
* Use of prophylactic headache medication within 28 days prior to week -4
* Unremitting headache lasting continuously throughout the 4-week baseline period
* Known or suspected Temporomandibular Disorders (TMD)
* Diagnosis of fibromyalgia
* Beck depression inventory score >24 at week-4
* Psychiatric problems that may have interfered with study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Allergan
Locations (2):
- Seattle, Washington, United States
- Markham, Ontario, Canada

REFERENCES:
- [Derived] Diener HC, Dodick DW, Lipton RB, Manack Adams A, DeGryse RE, Silberstein SD. Benefits Beyond Headache Days With OnabotulinumtoxinA Treatment: A Pooled PREEMPT Analysis. Pain Ther. 2020 Dec;9(2):683-694. doi: 10.1007/s40122-020-00198-w. Epub 2020 Oct 7. PMID 33026631
- [Derived] Silberstein SD, Diener HC, Dodick DW, Manack Adams A, DeGryse RE, Lipton RB. The Impact of OnabotulinumtoxinA vs. Placebo on Efficacy Outcomes in Headache Day Responder and Nonresponder Patients with Chronic Migraine. Pain Ther. 2020 Dec;9(2):695-707. doi: 10.1007/s40122-020-00199-9. Epub 2020 Oct 7. PMID 33026630
- [Derived] Dodick DW, Silberstein SD, Lipton RB, DeGryse RE, Adams AM, Diener HC. Early onset of effect of onabotulinumtoxinA for chronic migraine treatment: Analysis of PREEMPT data. Cephalalgia. 2019 Jul;39(8):945-956. doi: 10.1177/0333102418825382. Epub 2019 May 21. PMID 31112399
- [Derived] Silberstein SD, Dodick DW, Aurora SK, Diener HC, DeGryse RE, Lipton RB, Turkel CC. Per cent of patients with chronic migraine who responded per onabotulinumtoxinA treatment cycle: PREEMPT. J Neurol Neurosurg Psychiatry. 2015 Sep;86(9):996-1001. doi: 10.1136/jnnp-2013-307149. Epub 2014 Dec 12. PMID 25500317
- [Derived] Rendas-Baum R, Yang M, Varon SF, Bloudek LM, DeGryse RE, Kosinski M. Validation of the Headache Impact Test (HIT-6) in patients with chronic migraine. Health Qual Life Outcomes. 2014 Aug 1;12:117. doi: 10.1186/s12955-014-0117-0. PMID 25080874
- [Derived] Aurora SK, Winner P, Freeman MC, Spierings EL, Heiring JO, DeGryse RE, VanDenburgh AM, Nolan ME, Turkel CC. OnabotulinumtoxinA for treatment of chronic migraine: pooled analyses of the 56-week PREEMPT clinical program. Headache. 2011 Oct;51(9):1358-73. doi: 10.1111/j.1526-4610.2011.01990.x. Epub 2011 Aug 29. PMID 21883197
- [Derived] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038

RESULTS

PARTICIPANT FLOW:
Period: Double-Blind Phase (DB)
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Started | 341 | 338
Completed | 296 (Completed Week 24) | 295 (Completed Week 24)
Not Completed | 45 | 43
Period: Open-Label Phase (OL)
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Started | 285 (Number of DB Botulinum toxin type A patients who rolled into OL phase) | 286 (Number of DB Placebo patients who rolled into OL Phase)
Completed | 252 | 231
Not Completed | 33 | 55

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo (Saline) | Total
Number analyzed (Participants) | 341 | 338 | 679
Age, Customized [Number; unit: participants]
  < 40years | 144 | 128 | 272
  >= 40 years | 197 | 210 | 407
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 290 | 594
  Male | 37 | 48 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Headache Episodes
Description: Mean change from baseline in frequency (number) of headache episodes during the 28 day period ending with Week 24. Headache episode defined as patient-reported headache with a start and stop time indicating that the pain lasted >= 4 continuous hours.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Headache Episodes
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 341 | 338
Headache Episodes
  Baseline | 12.3 (5.23) | 13.4 (5.71)
  Change from Baseline at Week 24 | -5.2 (5.27) | -5.3 (5.85)

2. Secondary Outcome: Change in Frequency of Headache Days
Description: Mean change from baseline in frequency (number) of headache days during the 28 day period ending with Week 24. Headache day defined as a calendar day [00:00 to 23:59] for which the patient reported >= 4 continuous hours of headache
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Headache Days
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 341 | 338
Headache Days
  Baseline | 20.0 (3.73) | 19.8 (3.71)
  Change from Baseline at Week 24 | -7.8 (6.57) | -6.4 (6.69)

3. Secondary Outcome: Change in Frequency of Acute Headache Pain Medication Intakes
Description: Mean change from baseline in frequency (number) of acute headache pain medication intakes during the 28 day period ending with Week 24. Medication intakes defined as the number of times a patient took acute headache pain medication regardless of dose or type/number of medications taken at the same time.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Medication Intakes
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 341 | 338
Medication Intakes
  Baseline | 29.1 (19.27) | 30.4 (22.29)
  Change from Baseline at Week 24 | -10.3 (18.67) | -10.4 (18.54)

4. Secondary Outcome: Change in Frequency of Migraine/Probable Migraine Headache Days
Description: Mean change from baseline in frequency (number) of migraine/probable migraine headache days during the 28 day period ending with Week 24. Headache day defined as a calendar day with >= 4 continuous hours of headache meeting ICHD-II criteria for migraine or probable migraine.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Migraine/Probable Migraine Headache Days
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 341 | 338
Migraine/Probable Migraine Headache Days
  Baseline | 19.1 (4.04) | 19.1 (4.05)
  Change from Baseline at Week 24 | -7.6 (6.51) | -6.1 (6.78)

5. Secondary Outcome: Change in Frequency of Migraine/Probable Migraine Headache Episodes
Description: Mean change from baseline in frequency (number) of migraine/probable migraine headache episodes during the 28 day period ending with Week 24. Headache episode defined as patient-reported headache with a start and stop time indicating that the pain lasted >= 4 continuous hours and met ICHD-II criteria for migraine or probable migraine.
Time Frame: Baseline, Week 24
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Migraine/Prob Migraine Headache Episodes
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Number analyzed (Participants) | 341 | 338
Migraine/Prob Migraine Headache Episodes
  Baseline | 11.5 (5.06) | 12.7 (5.72)
  Change from Baseline at Week 24 | -4.8 (5.06) | -4.9 (5.74)

ADVERSE EVENTS:
Description: For SAEs/AEs, the Total # Participants at Risk for the Botulinum toxin type A arm includes ALL patients in the safety population who received Botulinum toxin type A in the Double-Blind and Open-Label phases. The total # Participants at Risk for the Placebo arm includes ONLY Double-blind Phase patients in the safety population who received Placebo.
Arm/Group | Botulinum Toxin Type A | Placebo (Saline)
Serious Adverse Events (participants affected / at risk) | 42/624 | 8/334
Other Adverse Events (participants affected / at risk) | 215/624 | 64/334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=624) | Placebo (Saline) (N=334)
Migraine (Nervous system disorders) | 4 | 0
Non-cardiac chest pain (General disorders) | 3 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Invertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Migraine without aura (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Parvovirus B19 serology positive (Investigations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Rocky mountain spotted fever (Infections and infestations) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Status migrainosus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal stoma complications (Injury, poisoning and procedural complications) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peridiverticular abscess (Infections and infestations) | 1 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=624) | Placebo (Saline) (N=334)
Neck pain (Musculoskeletal and connective tissue disorders) | 63 | 11
Sinusitis (Infections and infestations) | 46 | 17
Upper respiratory tract infection (Infections and infestations) | 37 | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 35 | 0
Nasopharyngitis (Infections and infestations) | 34 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.